CLINICAL TRIAL: NCT07037485
Title: The Predictive Value of Doppler Based Renal Ultrasound and Urinary Oxygen Tension for Prediction of Acute Kidney Injury After Open Heart Surgery
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Mohamed Badr Ali Badr, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Other Study IDs: 36265MD279/9/24
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Doppler-Based Renal Ultrasound; Urinary Oxygen Tension; Acute Kidney Injury; Open Heart Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing elective on-pump cardiac surgery
  Interventions: Other: Renal resistive index; Other: Renal Artery Pulsatility Index; Other: Urinary oxygen tension (PUO2)

INTERVENTIONS:
Other: Renal resistive index — It will be measured with ultrasound-Doppler using an abdominal curvilinear probe ultrasonography by two independent, trained sonographers (who will not be involved in patient care). After visualizing the kidney in ultrasound mode and checking for renal abnormalities, an arcuate or inter-lobar artery will be localized, and three successive Doppler measurements at different positions in the kidney (high, middle, and low) will be performed. The average value for each kidney will be taken.
  The renal resistive index will be calculated as follows:
  (systolic peak flow velocity - diastolic minimum flow velocity)/systolic peak flow velocity
Other: Renal Artery Pulsatility Index — It will be measured using an abdominal curvilinear probe ultrasonography by two independent, trained sonographers (who will not be involved in patient care). After visualizing the kidney, the interlobular artery will be located using color Doppler mode, and the velocity of the interlobular arteries will be assessed in one or two kidneys.
  The Renal Artery Pulsatility Index (RAPI) will be calculated as follows:
  RAPI = [(peak systolic velocity) - (end diastolic velocity)] /average velocity
Other: Urinary oxygen tension (PUO2) — Urinary oxygen tension (PUO2) will be measured preoperatively (baseline), postoperatively just after intensive care unit admission, 12 hours after surgery, and then once daily for 7 days.

SUMMARY:
This study aims to investigate the predictive value of Doppler-based renal ultrasound and urinary oxygen tension in the development of acute kidney injury after cardiac surgery.

DETAILED DESCRIPTION:
Cardiac surgery-associated acute kidney injury (CSA-AKI) is a complication following cardiac surgery occurring in 15-30% of patients. It is associated with increased morbidity and mortality as well as prolonged hospital stay and higher medical costs.

The renal artery pulsatility index (RAPI), which is determined using Doppler measurements, has been reported to detect patients with a high risk of AKI. Additionally, the renal resistance index (RRI), measured by Doppler ultrasound, can accurately predict the occurrence of AKI.

Urinary oxygen partial pressure in the bladder has been shown to decrease in the setting of sepsis, reduced renal blood flow, and decreased cardiac output.

ELIGIBILITY:
Inclusion Criteria:

* Age above 21 years.
* Both sexes.
* Undergoing elective on-pump cardiac surgery.

Exclusion Criteria:

* Patients with chronic kidney disease.
* Patients with any renal pathology or anatomic kidney abnormalities.
* Patients on renal replacement therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort observational study will be conducted at Tanta University Hospitals for a period of at least two years, from October 2024 to September 2026, pending approval from the institutional ethics committee.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of cases developed acute kidney injury | 7 days after the procedure
  Number of cases developed acute kidney injury as defined by KIDGO guidelines (serum creatinine ≥ 0.3 mg/dL from base line within 48 hours, or ≥1.5 fold within 7 days, or urine output <0.5 mL/kg/hour for six hours) in patients undergoing open heart surgery.

SECONDARY OUTCOMES:
Length of intensive care unit stay | 7 days after the procedure
  The length of stay in an Intensive Care Unit (ICU) is defined as the duration a patient spends in the ICU, typically measured from the time of admission to the ICU until the time of discharge.
Length of hospital stay | 7 days after the procedure
  Length of hospital stay will be measured from admission till discharge from hospital.
Need for renal replacement therapy | 7 days after the procedure
  Need for renal replacement therapy will be recorded.
Number of patients developed chronic kidney disease | 7 days after the procedure
  Number of patients developed chronic kidney disease will be recorded.
Mortality rate | 7 days after the procedure
  Mortality rate will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.